CLINICAL TRIAL: NCT07389083
Title: The Efficacy and Safety of the Supraglottic Oxygenation Via Nasotracheal Intubation Reduce the Incidence of Hypoxia in Patients Undergoing Sedated Fiberoptic Bronchoscopy.
Brief Title: The Efficacy and Safety of the Supraglottic Oxygenation Via Nasotracheal Intubation for Deep Sedation Fiberoptic Bronchoscopy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Principal Investigator, Yueying Zheng, Deputy Director of the Anesthesiology Department, First Affiliated Hospital of Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ZJU2025C180
Record Dates: First submitted 2025-12-31; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-11

CONDITIONS: Hypoxia; Pulmonary Nodule; Pulmonary Infection
Keywords: fiberoptic bronchoscopy; Hypoxia; Deep sedation; supine position; tongue-base fallback; supraglottic oxygenation
MeSH Terms: conditions — Hypoxia; Deception

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supraglottic oxygenation via nasotracheal catheterization Airway Group (Other): In this group, patients received supraglottic oxygen therapy via nasotracheal intubation.
  Interventions: Device: wire-reinforced tracheal tube

INTERVENTIONS:
Device: wire-reinforced tracheal tube — Supraglottic oxygen therapy delivered via wire-reinforced nasotracheal tube

SUMMARY:
Bronchoscopy is now widely used for the diagnosis and treatment of various respiratory diseases. However, the procedure is highly stimulating and provokes a strong stress response; because the airway is shared, patients are prone to hypoxia. With the growing emphasis on comfortable care, demand for anesthesia during bronchoscopy has increased. Deep sedation is the most common approach, but when administered in the supine position it often causes the tongue base to fall back. Both nasopharyngeal and oropharyngeal airways can relieve this obstruction, yet neither connects seamlessly to an oxygen supply line, resulting in insufficient oxygen delivery.We therefore replaced the nasopharyngeal airway with a wired endotracheal tube (size 4.0 or 4.5) inserted via the nose. This thinner tube couples easily to an oxygen line or ventilator circuit, partially relieves airway obstruction, and allows ample supraglottic oxygenation. The present study was designed to evaluate the feasibility and safety of this modified oxygen-delivery method in patients undergoing deep sedation for bronchoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing fiberoptic bronchoscopy under deep sedation.
* Written informed consent obtained from the patient or their legal representative.
* Clear understanding of, and voluntary participation in, the study, with informed-consent form signed by the patient or their legal representative.

Exclusion Criteria:

* Age < 18 years
* BMI > 30 kg/m²
* Previous history of abnormal recovery from anesthesia/surgery
* History of recurrent epistaxis, nasal bone fracture, nasal polyps, or sinus surgery
* Chronic use of opioid analgesics, benzodiazepine hypnotics, or antidepressant medications
* Known allergy to any of the anesthetic agents employed
* Anticipated difficult airway
* Increased intracranial pressure
* Active upper-respiratory-tract infection of the oral, nasal, or pharyngeal regions
* Severe cardiac insufficiency (functional capacity < 4 METs)
* Severe renal failure requiring dialysis prior to surgery
* Pre-operative oxygen saturation on room air < 92 %
* Any condition that, in the opinion of the investigator, renders the patient unsuitable for participation in this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-12-28 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
The incidence of hypoxia（75% ≤ SpO2 < 90% for <60 s） | Periprocedural

SECONDARY OUTCOMES:
The incidence of sub-clinical respiratory depression(90% ≤ SpO2 < 95%) | Periprocedural
The incidence of severe hypoxia(SpO2 < 75% or 75% ≤ SpO2 < 90% for ≥60 s) | Periprocedural

OTHER OUTCOMES:
To observe the incidence of adverse events according to the document from the World SIVA International Sedation Task Force(doi:10.1093/bja/aer407) in patients undergoing bronchoscopy under deep sedation | peri-anesthetic period

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol